CLINICAL TRIAL: NCT01594710
Title: Risk Factor Analysis for Developing Metabolic Syndrome in Korean Adults
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor, Korea University
Other Study IDs: KoreaHealth_MS
Record Dates: First submitted 2012-04-28; First posted 2012-05-09 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2014-04

CONDITIONS: Metabolic Syndrome, Atherosclerosis
MeSH Terms: conditions — Metabolic Syndrome; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Apparently Health People

SUMMARY:
In Asia, the prevalence of metabolic syndrome have been dramatically increased. Therefore, the investigators intend to the collect the blood sample, laboratory, anthropometric, and body composition parameters prospectively to examine the risk factors of metabolic syndrome. Furthermore, the investigators will collect the data of carotid IMT and branchial ankle pulse wave velocity to clarify the metabolic risk factors of atherosclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy people who underwent medical routine check up in Korea Health Promotion Center.
* age > 20 years

Exclusion Criteria:

* History of cardiovascular disease (myocardial infarction, unstable angina, stroke, or cardiovascular revascularization)
* Stage 2 hypertension
* Severe renal or hepatic disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Apparently healthy people who underwent medical routine check up in Korea University Helath Promotion Center.
Sampling Method: Probability Sample
Enrollment: 1800 (Actual)
Dates: Start 2012-02; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
The impact of various cardiovascular risk factors (inflammatory markers, hepatokines, adipokines, body composition parameters) for developing metabolic syndrome in prospective design | 36months

SECONDARY OUTCOMES:
The relationship of various cardiovascular risk factors (inflammatory markers, hepatokines, adipokines, body composition parameters) with metabolic syndrome and atherosclerosis measured by baPWV and carotid IMT in cross sectional design | 36months

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yoo HJ, Hwang SY, Choi JH, Lee HJ, Chung HS, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Association of leukocyte cell-derived chemotaxin 2 (LECT2) with NAFLD, metabolic syndrome, and atherosclerosis. PLoS One. 2017 Apr 4;12(4):e0174717. doi: 10.1371/journal.pone.0174717. eCollection 2017. PMID 28376109
- [Derived] Lee HJ, Hwang SY, Hong HC, Ryu JY, Seo JA, Kim SG, Kim NH, Choi DS, Baik SH, Choi KM, Yoo HJ. Waist-to-hip ratio is better at predicting subclinical atherosclerosis than body mass index and waist circumference in postmenopausal women. Maturitas. 2015 Mar;80(3):323-8. doi: 10.1016/j.maturitas.2014.12.015. Epub 2015 Jan 12. PMID 25631349
- [Derived] Yoo HJ, Hwang SY, Hong HC, Choi HY, Seo JA, Kim SG, Kim NH, Choi DS, Baik SH, Choi KM. Association of metabolically abnormal but normal weight (MANW) and metabolically healthy but obese (MHO) individuals with arterial stiffness and carotid atherosclerosis. Atherosclerosis. 2014 May;234(1):218-23. doi: 10.1016/j.atherosclerosis.2014.02.033. Epub 2014 Mar 16. PMID 24681911
- [Derived] Choi KM, Hwang SY, Hong HC, Choi HY, Yoo HJ, Youn BS, Baik SH, Seo HS. Implications of C1q/TNF-related protein-3 (CTRP-3) and progranulin in patients with acute coronary syndrome and stable angina pectoris. Cardiovasc Diabetol. 2014 Jan 13;13:14. doi: 10.1186/1475-2840-13-14. PMID 24417980
- [Derived] Hong HC, Hwang SY, Choi HY, Yoo HJ, Seo JA, Kim SG, Kim NH, Baik SH, Choi DS, Choi KM. Relationship between sarcopenia and nonalcoholic fatty liver disease: the Korean Sarcopenic Obesity Study. Hepatology. 2014 May;59(5):1772-8. doi: 10.1002/hep.26716. Epub 2014 Mar 24. PMID 23996808